CLINICAL TRIAL: NCT07268521
Title: A Multicenter Phase 2 Single-arm Proof-of-concept Trial Assessing the Efficacy and Safety of Obinutuzumab in the Treatment of Non-infectious Active Cryoglobulinemia Vasculitis Refractory or Intolerant to Rituximab
Acronym: CRYOBI
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP230848
Record Dates: First submitted 2025-11-18; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Cryoglobulinemic Vasculitis (CV)
Keywords: Cryoglobulinemic vasculitis (CV)
MeSH Terms: conditions — Cryoglobulinemia, Familial Mixed | interventions — obinutuzumab

STUDY DESIGN:
Intervention Model Description: multicenter open pilot phase 2 single arm prospective study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult patients with non-infectious active cryoglobulinemia vasculitis (Experimental)
  Interventions: Drug: Obinutuzumab

INTERVENTIONS:
Drug: Obinutuzumab — Obinutuzumab will be administered intravenously at 1000 milligrams (mg) at week 0 and week 2

SUMMARY:
Cryoglobulinemic vasculitis (CV) is a rare life threatening systemic immune-complex-mediated vasculitic syndrome. Symptoms range from arthralgia, purpura to more severe manifestations such as peripheral neuropathy, glomerulonephritis, and skin necrosis.1 CV is associated with significant morbidity and mortality. The management of non-infectious mixed CV is currently based on steroids, and anti-CD20 monoclonal antibody Rituximab (RTX). Infectious complications of immunosuppressants (IS) remain the main cause of death in CV. During the last decade, studies reported efficacy of RTX in patients with CV in 65-70% of patients as compared to 30% for other IS (azathioprine…). However, CV relapse is noted in up to 40% patients within few days to 19 months after the last RTX infusion2. Following RTX, serum levels of B lymphocyte stimulator (BLyS) significantly increased and may favour the survival of autoreactive B cell clones and relapses of CV. A recent study has shown that RTX does not reset defective early B cell tolerance checkpoints. Incomplete B cell depletion following treatment with RTX may be associated with poor clinical response.

Moreover, some patients develop a serum sickness reaction to RTX that contraindicate further use of the medication2. Thus, there are important therapeutic unmet needs in CV patients that are refractory or intolerant to RTX.

Obinutuzumab (OBZ) is a type II anti-CD20 monoclonal antibody with a glycomodified Fc, approved in 2013 for the treatment of chronic lymphocytic leukemia. Reddy et al. found that OBZ was at least 2-fold more efficient than RTX at inducing B-cell cytotoxicity in in vitro whole blood assays of patients with rheumatoid arthritis and systemic lupus erythematosus. In lupus nephritis, OBZ resulted in increased complete and partial renal responses compared with placebo when added to mycophenolate mofetil and steroids for the treatment of lupus nephritis. There is a strong rationale for using OBZ in CV. OBZ is currently used off label in CV patients intolerant to RTX and case reports pointed out its effectiveness in CV4.5. CRYOBI is the first prospective multicenter phase 2 proof-of-concept trial assessing efficacy of OBZ in CV refractory or intolerant to RTX.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Written informed consent
3. Active mixed cryoglobulinemia vasculitis defined by:

   * a clinically active vasculitis signs with skin, joint, renal, peripheral nerve, central neurological, digestive, pulmonary
   * and/or cardiac involvement,
   * and history of positive cryoglobulinemia and/or positive Rheumatoid factor associated with low C4 complement level, and/or a monoclonal component (IgM Kappa) and/or a histological proof of vasculitis in the affected organs
4. Refractory or intolerant to Rituximab.

   Refractory patients are defined as any of the following after a standard rituximab regimen (375 mg/m² IV weekly for 4 consecutive weeks):
   * No measurable improvement within 4-6 weeks of initiation,
   * OR <50% improvement in the number or severity of affected organ systems at 12 weeks, or
   * OR Persistent baseline manifestations without remission or significant improvement for >12 weeks.

   Improvement: A measurable positive change in the clinical signs, symptoms, and/or functional status of the affected organ(s), compared to baseline, as assessed using the organ-specific criteria below, without fulfilling full remission requirements.

   Remission: Complete disappearance of all baseline symptoms and objective abnormalities in the affected organ(s), as defined below:

   "CRYOBI " protocol, version v1-2 of 26/08/2025 10/68 This document is the property of DRCI/AP-HP. All reproduction is strictly prohibited. Version 4.0 dated 31/05/2019
   * The skin and articular remissions are evaluated clinically (disappearance of purpura and ulcers, disappearance of arthritis, disappearance of the skin necrosis).
   * Renal remission is evaluated biologically (proteinuria <0.5g/24h or proteinuria/creatininuria <50 mg/mmol), and improvement of GFR >20% if GFR <60 mL/min/1.73 m2 at diagnosis or glomerular filtration rate ≥60ml/min/1.73m² if GFR ≥ 60 mL/min1.73 m2 at diagnosis
   * Peripheral Neurological remission is evaluated clinically (any improvement of pains and paresthesia by visual analogue scales, any stabilization or improvement of muscular testing in case of motor impairment at baseline) and electrophysiologically (stabilization or improvement of electromyogram abnormalities compared to baseline).
   * Central Neurological remission is evaluated clinically (no new neurological symptoms and stabilization or improvement of the initial presentation) and radiologically (Cerebral MRI showing no new lesions and no contrast enhancement of the initial lesions, or regression of the initial lesion)
   * Digestive remission is evaluated clinically (resolution of abdominal pain and other gastrointestinal symptoms), and by endoscopy (resolution of potential gastrointestinal lesions seen at baseline) and/or by CT scan (resolution of any abnormalities found on baseline imaging). Complete remission of all baseline abnormalities is required to define digestive remission.
   * Cardiac remission is evaluated clinically (resolution of chest pains and other cardiac events), and biologically (normalization of myocardial enzymes) and radiologically (no late gadolinium enhancement on cardiac MRI). Complete remission of all baseline abnormalities is required to define cardiac remission.

   Pulmonary remission: complete regression of the initial symptoms with no new radiological lesions and regression of all the initial lesions.

   Intolerant: Patients who experienced treatment-limiting adverse events or toxicity that required discontinuation of rituximab, despite dose modification or supportive care.
5. HIV negative serology within 3 months prior inclusion
6. Negative HBs Ag test within 3 months prior inclusion. (In case of negative AgHBs and positive HBc Ab test, HBV DNA test must be negative; AND Hepatitis B surveillance should be started (monthly HBsAg and HBV DNA testing for the duration of the study treatment and at least every 12 weeks after treatment is discontinued for the duration of study treatment. In addition, antiviral prophylaxis should be started before the first administration of the study treatment and continued until 12 months after completion of study treatment)
7. HCV negative serology or negative HCV RNA if positive HCV serology within 3 months before inclusion
8. Affiliated to National French social security system (registered or being a beneficiary of such a scheme). Patients with AME are eligible

Exclusion Criteria:

1. Vasculitis unrelated to cryoglobulinemia
2. Non-active cryoglobulinemia vasculitis
3. Treatment with cyclophosphamide or Belimumab within 3 months prior to inclusion
4. Malignant neoplasm within the last 5 years other than carcinoma in situ of the cervix or excised basal cell, squamous cell carcinoma of the skin and low-grade hemopathy with no indication for a specific treatment.

   "CRYOBI " protocol, version v1-2 of 26/08/2025 11/68 This document is the property of DRCI/AP-HP. All reproduction is strictly prohibited. Version 4.0 dated 31/05/2019 Carcinoma in situ of the cervix and squamous cell carcinoma of the skin should have been adequately treated before inclusion in the study.
5. Active tuberculosis, pneumocystis, cytomegalovirus or any active infection not adequately managed or considered a risk by the investigator
6. Have a history of an anaphylactic reaction to parenteral administration of Obitunuzumab
7. Unstable or high-risk cardiac conditions, e.g., recent (<6 months) myocardial infarction or unstable angina, decompensated (NYHA III-IV) heart failure, clinically significant uncontrolled arrhythmias, or any cardiac condition that, in the investigator's judgment, poses an unacceptable risk with obinutuzumab infusion
8. Pregnant or breastfeeding women, or desire to become pregnant within 30 months All women of childbearing potential (WOCBP) are required to have a negative pregnancy test before treatment and must agree to maintain highly effective contraception by practicing abstinence or by using an effective method of birth control from the date of consent until 18 months after the last obinutuzumab infusion: Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (Oral, Intravaginal, Transdermal); Progestogen-only hormonal contraception associated with inhibition of ovulation (Oral, Injectable, Implantable); Intrauterine device (IUD); Intrauterine hormone-releasing system (IUS); Bilateral tubal occlusion; Vasectomised partner
9. Neutrophils < 1000/mm3 or Platelets < 50000/mm3
10. Live vaccines within 30 days prior inclusion
11. Patients under guardianship or curatorship and protected adults or unable to consent
12. Progressive multifocal leukoencephalopathy
13. Participation to another interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Complete Clinical Response | At 6 months
  Remission of all affected organs involved at baseline and with corticosteroid withdrawal in the absence of severe clinical relapse

SECONDARY OUTCOMES:
Frequency of adverse clinical events | At 12 weeks
  Frequency and severity of adverse clinical events
Frequency of adverse clinical events | At 24 weeks
  Frequency and severity of adverse clinical events
Frequency of adverse clinical events | At 48 weeks
  Frequency and severity of adverse clinical events
Rates of patients with complete clinical response with corticosteroid withdrawal (prednisone at 0 mg/day), partial response, and no clinical response | At 12 weeks
Rates of patients with complete clinical response with corticosteroid withdrawal (prednisone at 0 mg/day), partial response, and no clinical response | At 24 weeks
Rates of patients with complete clinical response with corticosteroid withdrawal (prednisone at 0 mg/day), partial response, and no clinical response | At 48 weeks
Rate of patients with complete renal remission | At 12 weeks
  Defined as proteinuria < 0.5g/24h or proteinuria/creatininuria < 50 mg/mmol, and improvement of GFR > 20% if GFR < 60 mL/min/1.73 m² at diagnosis or GFR > 60 mL/min/1.73m² if GFR ≥ 60ml/min/1.73m² at diagnosis.
Rate of patients with complete renal remission | At 24 weeks
  Defined as proteinuria < 0.5g/24h or proteinuria/creatininuria < 50 mg/mmol, and improvement of GFR > 20% if GFR < 60 mL/min/1.73 m² at diagnosis or GFR > 60 mL/min/1.73m² if GFR ≥ 60ml/min/1.73m² at diagnosis.
Rate of patients with complete renal remission | At 48 weeks
  Defined as proteinuria < 0.5g/24h or proteinuria/creatininuria < 50 mg/mmol, and improvement of GFR > 20% if GFR < 60 mL/min/1.73 m² at diagnosis or GFR > 60 mL/min/1.73m² if GFR ≥ 60ml/min/1.73m² at diagnosis.
Rate of patients without cryoglobulinemia | At 12 weeks
Rate of patients without cryoglobulinemia | At 24 weeks
Rate of patients without cryoglobulinemia | At 48 weeks
Rate of patients without rheumatoid factor activity | At 12 weeks
Rate of patients without rheumatoid factor activity | At 24 weeks
Rate of patients without rheumatoid factor activity | At 48 weeks
Rate of patients with normal C4 complement level | At week 12
Rate of patients with normal C4 complement level | At week 24
Rate of patients with normal C4 complement level | At week 48
Rate of patients with early treatment failure | At week 4
  Defined as the absence of clinical response
Cumulative incidence of clinical relapse (severe or non-severe) | Up to 144 weeks
  Defined by reappearance of a manifestation attributable to cryoglobulinemia vasculitis
Cumulative incidence of severe clinical relapse | Up to 144 weeks
  A severe relapse is defined by the appearance or reappearance of one of the following signs:
  * Extensive skin necrosis with loss of substance
  * Specific cardiac involvement of vasculitis (documented by EKG, troponin and/or MRI)
  * Specific digestive impairment of vasculitis (documented by imaging and/or endoscopy)
  * Affection of the central nervous system specific to vasculitis (documented by cerebral MRI)
  * Multiple mononeuropathy clinically defined by asymmetrical motor impairment of 2 or more nerve trunks. (Documented by electromyogram)
  * Severe renal impairment defined as a doubling of creatinine levels from the usual value or a glomerular filtration rate according to CKD-EPI of less than 30 ml/min/1.73m2 in the absence of prior history of creatinine levels)
Cumulative incidence of mild or moderate clinical relapse | Up to 144 weeks
  * Appearance or reappearance of purpura
  * Arthritis
  * Sensory neuropathy documented by electromyogram
  * Glomerulonephritis (proteinuria>1g/24h after excluding other causes of proteinuria)
Cumulative dose of prednisone | At week 24
Cumulative dose of prednisone | At 48 weeks
Birmingham Vasculitis Activity Score (BVAS) activity score variation | Up to 12 weeks
  Standardized clinical tool used to quantify disease activity. It varies from 0 to 63. The higher the BVAS, the more active and severe the vasculitis.
  Variation assessed from baseline
Birmingham Vasculitis Activity Score (BVAS) activity score variation | Up to 24 weeks
  Standardized clinical tool used to quantify disease activity. It varies from 0 to 63. The higher the BVAS, the more active and severe the vasculitis.
  Variation assessed from baseline
Birmingham Vasculitis Activity Score (BVAS) activity score variation | Up to 48 weeks
  Standardized clinical tool used to quantify disease activity. It varies from 0 to 63. The higher the BVAS, the more active and severe the vasculitis.
  Variation assessed from baseline
Variation in physical summary components of score SF-36 | Up to 24 weeks
  SF-36 assesses overall health-related quality of life across multiple domains. Each domain is scored from 0 to 100. 0 = worst possible health status 100 = best possible health status It is assessed from baseline.
Variation in physical summary components of score SF-36 | Up to 48 weeks
  SF-36 assesses overall health-related quality of life across multiple domains. Each domain is scored from 0 to 100. 0 = worst possible health status 100 = best possible health status It is assessed from baseline.
Variation in mental summary components of score SF-36 | Up to 24 weeks
  SF-36 assesses overall health-related quality of life across multiple domains. Each domain is scored from 0 to 100. 0 = worst possible health status 100 = best possible health status It is assessed from baseline.
Variation in mental summary components of score SF-36 | Up to 48 weeks
  SF-36 assesses overall health-related quality of life across multiple domains. Each domain is scored from 0 to 100. 0 = worst possible health status 100 = best possible health status It is assessed from baseline.
Cumulative incidence of infections (severe or non-severe) | Up to 48 weeks
  From baseline
Cumulative incidence of severe infections | Up to 48 weeks
  From baseline
  Severe infection defined by:
  * Tuberculosis, pneumocystis, or cytomegalovirus,
  * Leading to hospitalization
  * Leading to life threatening or death
    - Progressive multifocal leukoencephalopathy.
  * If PML is confirmed, study agent should be discontinued and consideration should be given to stopping immunosuppressant therapy.
    * Neoplasia
    * Serious Hypersensitivity or Infusion Reactions ≥ grade 3 CTCAE
    * Clinically significant, potentially life-threatening (Grade 4) adverse event (AE) that the investigator believes is definitely, possibly or probably related to study agent.
Cumulative incidence of non-severe infections | Up to 48 weeks
  From baseline Infections that do not meet the definition of a "severe infection"
Cumulative incidence of non-infectious complications (cancer, lymphoma, cardiovascular event: stroke, myocardial infarction, renal replacement, …) | Up to 48 weeks
  From baseline
Variation of gammaglobulin and of CD19+ B cells levels | Up to 12 weeks
  From baseline
Variation of gammaglobulin levels | Up to 24 weeks
  From baseline
Variation of gammaglobulin levels | Up to 48 weeks
  From baseline
Overall survival | Up to 144 weeks
  From baseline
Variation of CD19+ B cells levels | Up to 24 weeks
  From baseline
Variation of CD19+ B cells levels | Up to 48 weeks
  From baseline

IPD SHARING:
Plan to Share IPD: Undecided